CLINICAL TRIAL: NCT05770388
Title: Development and Evaluation of a Digital Technology-based Programme for Detecting Suicidal Risk and Promoting Help-seeking Among University Students: a Feasibility Study (Pilot RCT)
Brief Title: App-based Intervention to Promote Mental Health Help-seeking Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: University Diego Portales (Other); Millennium Nucleus to Improve the Mental Health of Adolescents and Youths (Imhay), ANID - NCS2021_081 (Unknown); Millennium Institute on Immunology and Immunotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONDECYT Postdoctorado 3200944
Record Dates: First submitted 2023-01-30; First posted 2023-03-15 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-08

CONDITIONS: Suicidal Ideation; Suicidal Behavior
Keywords: Suicide Prevention; Help-Seeking Behavior; App-based Intervention; University Students
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention; Help-Seeking Behavior | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants will receive a brief contact intervention (via phone call or chat) in which a clinical psychologist will assess their general mental health status and level of suicidal risk, and will provide an intervention based on the principles of motivational interviewing and psycho-educational information along with a list of mental health services available within and outside the University. Participants will also receive instructions on how to download and use a mobile app.
  Interventions: Device: App Take Care of Your Mood
- Intervention Group (Experimental): Participants will receive a brief contact intervention (via phone call or chat) in which a clinical psychologist will assess their mental health status and level of suicidal risk and will provide an intervention based on the principles of motivational interviewing and psycho-educational information along with a list of mental health services available within and outside the University. Participants will also receive instructions on how to download and use a mobile app. Additionally, participants will also receive reminder messages (by email and chat) encouraging them to use the app and to request a counseling session (via phone call, videoconference or chat) with a clinical psychologist if they think it is necessary. After two months, this group will receive a new contact with a clinical psychologist via phone call or chat. In this contact, mood and level of suicidal risk will be assessed, and participants will be encouraged to seek mental health help if they have not already done so.
  Interventions: Device: App Take Care of Your Mood; Behavioral: Reminder messages and counseling

INTERVENTIONS:
Device: App Take Care of Your Mood — The app provides psychoeducational information, contains several thematic modules (mindfulness, emotional regulation, healthy lifestyle habits, safety plan for crisis management, among others), allows mood monitoring, contains motivational messages and videos aimed at promoting help-seeking in mental health, and information on available support services.
Behavioral: Reminder messages and counseling — Participants receive reminder messages (by email and chat) encouraging them to use the app and to request a counseling session (via phone call, videoconference or chat) with a clinical psychologist if they think it is necessary.
  Arms: Intervention Group

SUMMARY:
It is estimated that approximately one in three university students has a mental health problem and between 5-10% have active suicidal ideation. Most college students do not receive professional treatment, which has been associated with structural and attitudinal barriers to help-seeking. Given that young people regularly use the internet to seek information about health problems, internet and digital technology-based interventions could represent an effective approach to overcome attitudinal barriers.

The goal of this study is to evaluate the feasibility of a mobile app-based intervention for the promotion of help-seeking in mental health services for university students at risk of suicide. The main questions it aims to answer are:

* Is it feasible to implement a mobile app-based intervention for the promotion of mental health help-seeking in a university context?
* Is it possible to increase the likelihood of help-seeking in mental health services among university students at risk of suicide through an app-based intervention?

Participants will receive a brief contact intervention (via phone call or chat) where they will be assessed by a clinical psychologist, receive information on available support services and instructions to download and use a mobile app called "Take Care of Your Mood". In addition, the participants can request a counseling session with a clinical psychologist. Participants will also receive reminder messages (by email and chat) motivating them to use the app or request a counseling session with a psychologist if they deem it necessary.

Researchers will compare this intervention with a brief contact intervention (control group) where participants will be assessed by a clinical psychologist, will receive instructions to download and use the app, but will not receive reminder messages or be able to access a counseling session with a psychologist.

ELIGIBILITY:
Inclusion Criteria:

* University students who have completed the Longitudinal Survey of University Student Mental Health (ELSAM), based on The WHO World Mental Health International College Student (WMH-ICS) initiative
* Suicidal ideation during the last 12 months
* Have access to Internet, email and Smartphone
* Agree to participate in the research through informed consent.

Exclusion Criteria:

* Currently undergoing mental health treatment (psychological or psychiatric)
* High suicidal risk during the last 30 days and/or 3 months [answer "yes" to questions 4 and 5 (last 30 days) and/or question 6 (last 3 months) of the C-SSRS]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Response, drop-out and adherence rates | 3 months post-randomization
  Data will be collected on the number of eligible individuals and those who enter the study. The response rate of participants and the adherence and dropout levels of participants during follow-up will also be evaluated.
Acceptance | 3 months post-randomization
  Acceptance will be assessed through 7 questions on perceived usefulness and relevance of the intervention, degree of engagement and participation, among others. The responses are made in a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate more acceptance of the program.
User Satisfaction | 3 months post-randomization
  Semi-structured interviews (n=15) will be conducted to explore participants' experience, evaluation of the app content, and opinions on potential changes to be included in the intervention.
User Experience | 3 months post-randomization
  The Standardized User Experience Percentile Rank Questionnaire for Mobile Apps (SUPR-Qm) will be used. The SUPR-Qm is a 16-item instrument that assesses a user's experience of a mobile application. The questionnaire has 16 items with responses on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree). Higher scores indicate a better evaluation of the app.

SECONDARY OUTCOMES:
Willingness to change | 3 months post-randomization
  Participants will answer the following question: "How would you rate your willingness or readiness to change emotional problems you may be having right now?" Answers can range from 1 ("I don't have any problems that need to change") to 5 ("I had a problem, but I have done something about it and things are going better now"). A higher score indicates a greater willingness to change.
Intention to help-seeking | 3 months post-randomization
  Participants will answer the following question: "Within the next 30 days, how likely do you think it is that you will seek help from a mental health service?" (1=very likely and 5=not at all likely). A lower score indicates a higher likelihood of seeking mental health help.
Access to treatment | 3 and 6 months post-randomization
  It will be assessed on the basis of a question on the use of mental health services (counselling, psychotherapy, pharmacotherapy or other) during the last 3 months (1=Yes, 2=No).
Barriers to accessing treatment | 3 months post-randomization
  It will be assessed on the basis of the "Seeking treatment" section of The WHO World Mental Health International College Student (WMH-ICS) Initiative questionnaire, which contains 10 items aimed at assessing attitudes towards seeking help and barriers to accessing treatment (Ebert et al. 2019). Responses to each item can range from 1 (very important) to 5 (not important).
Suicidal risk | 3 months post-randomization
  The Columbia Suicide Severity Rating Scale (C-SSRS) is an interviewer-rated measure of suicidal thoughts and behaviors. The abbreviated version of the scale contains 6 questions and classifies people into three groups (no risk or slight risk, moderate risk, high risk). Scores can range from 0 to 6. Higher scores represent a higher risk of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Jiménez-Molina, PhD, Principal Investigator — University Diego Portales
Locations (1):
- Álvaro Jiménez-Molina, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auerbach RP, Mortier P, Bruffaerts R, Alonso J, Benjet C, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Murray E, Nock MK, Pinder-Amaker S, Sampson NA, Stein DJ, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. J Abnorm Psychol. 2018 Oct;127(7):623-638. doi: 10.1037/abn0000362. Epub 2018 Sep 13. PMID 30211576
- [Background] Bruffaerts R, Mortier P, Auerbach RP, Alonso J, Hermosillo De la Torre AE, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Stein DJ, Ennis E, Nock MK, Pinder-Amaker S, Sampson NA, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. Lifetime and 12-month treatment for mental disorders and suicidal thoughts and behaviors among first year college students. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1764. doi: 10.1002/mpr.1764. Epub 2019 Jan 20. PMID 30663193
- [Background] Jiménez-Molina A, Franco P, Mac-Ginty S, and Martínez V (2023) Internet-based interventions for prevention and early treatment of depression in higher education students. En Martínez V. y Miranda C. (eds) Prevention and early treatment of depression through the life course. Springer, 97-119. https://doi.org/10.1007/978-3-031-13029-8_6
- [Background] Ebert DD, Franke M, Kahlke F, Kuchler AM, Bruffaerts R, Mortier P, Karyotaki E, Alonso J, Cuijpers P, Berking M, Auerbach RP, Kessler RC, Baumeister H; WHO World Mental Health - International College Student collaborators. Increasing intentions to use mental health services among university students. Results of a pilot randomized controlled trial within the World Health Organization's World Mental Health International College Student Initiative. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1754. doi: 10.1002/mpr.1754. Epub 2018 Nov 20. PMID 30456814
- [Background] Mortier P, Cuijpers P, Kiekens G, Auerbach RP, Demyttenaere K, Green JG, Kessler RC, Nock MK, Bruffaerts R. The prevalence of suicidal thoughts and behaviours among college students: a meta-analysis. Psychol Med. 2018 Mar;48(4):554-565. doi: 10.1017/S0033291717002215. Epub 2017 Aug 14. PMID 28805169
- [Background] Martinez V, Espinosa-Duque D, Jimenez-Molina A, Rojas G, Vohringer PA, Fernandez-Arcila M, Luttges C, Irarrazaval M, Bauer S, Moessner M. Feasibility and Acceptability of "Cuida tu Animo" (Take Care of Your Mood): An Internet-Based Program for Prevention and Early Intervention of Adolescent Depression in Chile and Colombia. Int J Environ Res Public Health. 2021 Sep 13;18(18):9628. doi: 10.3390/ijerph18189628. PMID 34574553